CLINICAL TRIAL: NCT04979299
Title: Assessment of Depression in the Elderly : a Bias Related to the Stigmatisation of Patients Presenting in Wheelchairs
Brief Title: Assessment of Depression (iCGI) in Older People, According to Their Presentation in a Wheelchair or an Ordinary Chair.
Acronym: WHEELDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Center Guillaume Régnier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC21_01GR_WHEELDEP
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Depression in Old Age
Keywords: elderly depression; stigma; iCGI
MeSH Terms: conditions — Social Stigma | interventions — Wheelchairs

STUDY DESIGN:
Intervention Model Description: We procede in a randomization 1:1, stratified by site. In one group, patients will be seated in a wheelchair and in the second group, patients will be seated in an regular chair. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes (SNOSE).
Who Masked: Outcomes Assessor
Masking Description: Participants included in the wheelchair group settle into a hospital wheelchair. The wheelchair comes from a batch of two, without specific brand, standard color.
  The videos are showed to 10 different psychiatrists whom each proceed to 10 iCGI rating assessments, after receiving methodological informations.
  The psychiatrists are blinded evaluators. They are not aware of the objective of the study focusing on the impact of the wheelchair. They will be decepted with the information that the study aim to evaluate the iCGI, as a new version of the CGI with elderly patients (we will procede to a feedback afterward).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wheelchair group (Experimental): Patients included in the " wheelchair " group will be asked to sit in a wheelchair during the interview;
  Interventions: Other: Wheelchair
- Control group (No Intervention): Patients included in the control group will sit in a regular chair during the interview.

INTERVENTIONS:
Other: Wheelchair — Patient will be asked to sit in a wheelchair, and a 5-minute video recording of spontaneous speech capturing the semi-structured iCGI interview is made.
  Arms: wheelchair group

SUMMARY:
This study aims to test for a " wheelchair effect ", as a potential impact of stigma, during the evaluation of clinical global impression of depression.Elderly patients will be asked to sit in a wheelchair, or in a regular chair during recording a 5 minute video of spontaneous speech collected the iCGI semi-structured interview.

The videos are showed to 10 different psychiatrists whom each proceed to 10 iCGI rating assessments.The psychiatrists are blinded evaluators. They are not aware of the real objective of the study.

DETAILED DESCRIPTION:
This is a multicentric, randomized study of depression severity assessments (by iCGI) for wheelchair sitting elderly patients versus regular chair sitting elderly patients.The iCGI is a validated scale to assess depression severity through 5 min videos viewing of semi-structured interviews. The frame of the interviews is made to obtain the material provided by the patients expected to facilitate the formation of an "impression", an empathetic feeling, based on phenomenological concepts. The clinical interview is close to day-to-day clinical practice.

Patients are randomized (1:1) into 2 groups: "wheelchair" group and control group.

After randomization, a 5-minute video of spontaneous speech collecting the semi-structured iCGI interview is recorded.

These videos will square the participant's face, torso, and thighs, with a ¾ angle, in order to visualise the patient and the chair he is sitting in. The face will not be blurred in order to access non his non-verbal communication.

The videos are viewed by 10 different psychiatrists whom each proceed to 10 iCGI rating assessments, The psychiatrists are blinded evaluators. They are not aware of the objective of the study focusing on the impact of the wheelchair. They will be decepted with the information that the study aim to evaluate the iCGI, as a new version of the CGI with elderly patients.

The 10 videos each psychiatrist have to assess are randomly selected following the next rules :

* Un unbalanced number of wheelchair and regular chair videos, so as they don't guess the study directly focuses on the wheelchair.
* The wheelchair/regular chair video ratio is 7/3 or 3/7 for each psychiatrist.
* Each video is visualised once by one psychiatrist. Our objective is to highlight an assessment bias related to physical disability in depression in the elderly with the aim of improving the practices of all professionals involved.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised or ambulatory patients
* Suffering mild to severe depression, according to PHQ-9 (Patient Health Questionnaire-9) score ⩾ 5 [11].
* Ability to understand the protocol.
* Signed consent of the participant regarding the given information.
* Subscription to the social security system.

Exclusion Criteria:

* Walking disability (including walking with human help required).
* Severe cognitive impairment diagnosed with MMSE (Mini Mental State Examination) score <18 within the last three months.
* Historical or current schizophrenia diagnosis recorded on the medical file.
* Historical or current neurological disease recorded on the medical file : Neurodegenerative disorders, stroke, epilepsy.
* Patients under guardianship or trusteeship.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
psychiatrists' assessment of depression severity with the iCGI scale | after including all patients in the study, up to 24 month
  The iCGI is a validated scale to assess depression severity through 5 min videos viewing of semi-structured interviews. We will compare the iCGI in the " wheelchair " group and the control group. Analyzes will be based on each group's mean score.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel RG ROBERT, MD, Principal Investigator — Centre Hospitalier Guillaume Régnier
Locations (2):
- France (2):
  - EPSM Saint Avé, Saint-Avé, Brittany Region
  - Centre Hospitalier Guillaume Regnier, Rennes, Ile Et Vilaine

IPD SHARING:
Plan to Share IPD: Yes
Data about study protocol and clinical information will be available on request from other researchers.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be availablefrom the moment a scientific publication is accepted to five years later.
Access Criteria: acces to data will be granted to researchers aiming to perform another analysis or to review the topic, or to perform a meta-analysis.

REFERENCES:
- [Background] Krendl AC, Kensinger EA, Ambady N. How does the brain regulate negative bias to stigma? Soc Cogn Affect Neurosci. 2012 Aug;7(6):715-26. doi: 10.1093/scan/nsr046. Epub 2011 Sep 5. PMID 21896496
- [Background] Henderson C, Noblett J, Parke H, Clement S, Caffrey A, Gale-Grant O, Schulze B, Druss B, Thornicroft G. Mental health-related stigma in health care and mental health-care settings. Lancet Psychiatry. 2014 Nov;1(6):467-82. doi: 10.1016/S2215-0366(14)00023-6. Epub 2014 Nov 5. PMID 26361202
- [Background] MacDonald ML, Butler AK. Reversal of helplessness: producing walking behavior in nursing home wheelchair residents using behavior modification procedures. J Gerontol. 1974 Jan;29(1):97-101. doi: 10.1093/geronj/29.1.97. No abstract available. PMID 4809670
- [Background] Delmas H, Batail JM, Falissard B, Robert G, Range M, Brousse S, Soulabaille J, Drapier D, Naudet F. A randomised cross-over study assessing the "blue pyjama syndrome" in major depressive episode. Sci Rep. 2017 Jun 1;7(1):2629. doi: 10.1038/s41598-017-02411-x. PMID 28572626
- [Background] Kadouri A, Corruble E, Falissard B. The improved Clinical Global Impression Scale (iCGI): development and validation in depression. BMC Psychiatry. 2007 Feb 6;7:7. doi: 10.1186/1471-244X-7-7. PMID 17284321
- [Background] Laux G; VIVALDI Study Group. The antidepressant agomelatine in daily practice: results of the non-interventional study VIVALDI. Pharmacopsychiatry. 2012 Nov;45(7):284-91. doi: 10.1055/s-0032-1309003. Epub 2012 May 16. PMID 22592503
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941